CLINICAL TRIAL: NCT04253288
Title: The French Registry Of Morbidity And Mortality Reviews (MMR) Meetings: Prospective Registration Of Clinical, Dosimetric And Individual Biological Radiosensitivity Data Of Patients With Severe Radiation Toxicity (PROUST STUDY)
Brief Title: Prospective Registration of mOrbidity and Mortality, individUal radioSensitivity and Radiation Technique (PROUST)
Acronym: PROUST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: K160101J
Record Dates: First submitted 2020-01-06; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2019-11

CONDITIONS: Radiotherapy
Keywords: MMR; Radiation toxicity; Radiosensitivity; Late effects
MeSH Terms: conditions — Radiation Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with severe radiation toxicity (Other): Patients who received radiotherapy and developed abnormal radiation-induced toxicity
  Interventions: Other: Morbidity Mortality Review (MMR)

INTERVENTIONS:
Other: Morbidity Mortality Review (MMR) — * Standardization of Morbidity Mortality Review (MMR) in radiotherapy centers
  * National database from MMR board meetings which include clinical , radiation technique and biological parameters of intrinsic radiosensitivity of patients
  Other Names: National database from MMR

SUMMARY:
Background: Recently, an increasing international interest has arisen in using morbidity and mortality rates to monitor the quality of hospital cares (1, 2). Many hospitals have integrated the morbidity and mortality review (MMR) meetings into their governance processes, by making them mandatory and more accountable for taking corrective action (3-5).

Quality of radiotherapy (RT) delivery is highly operator dependent. The operator is a team of professionals including radiation oncologists, planning dosimetrists, physicists and technicians. Because of this complex, multi-step process, there is margin for error, which may affect outcomes and toxicity. Some deviations may have minimal effects on outcome, while others may have a profound effect and compromise long-term results. For the morbidity after RT, MMR is identified as one of the most adapted process to highlight whether and how these meetings provide assurance within the organizations' governance processes in radiation departments.

In France, many teams have not reached a formalized procedure for a systematic MMR. Furthermore, implementation of MMR in RT departments is very heterogeneous and not always meets the criteria defined by the Health Authorities (HAS) (6).

Systemic analysis conducted during the MMR is a comprehensive analysis of the situation, taking into account all technical and human elements. The diagnosis and type of morbidity depends on the irradiated volume, the dose delivered to the organ at risk and the individual radiosensitivity.

Follow-up after RT is important to evaluate outcome results and late toxicity. In general, late effects consist of tissue fibrosis and vascular damage, which can result in cosmetic and functional deterioration. Some of the radiation-induced sequelea may require particular management including hospitalization (lung fibrosis, gastro-intestinal and genito-urinary toxicities,..), while for other ones, only local treatments are needed (mucosal toxicity, skin fibrosis…). The challenge for clinicians in the frame of the MMR is to make sure that there is no controversy about the delivered RT quality and investigate other potential causes such as particular intrinsic radiosensitivity of the patient for a given standard treatment.

DETAILED DESCRIPTION:
The study consist of a prospective registration in a dedicated database (PROUST) of severe radiation toxicity that aims to implement MMR procedure in the French radiotherapy departments.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients who received RT alone or associated to other anti-cancer treatments
* Significant and durable toxicity grade > 3 whatever the organs concerned by radiation exposure
* Completion of baseline clinical and dosimetric data collection
* Patients with no psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
* Signed informed consent to participate in the study must be obtained from patients after they have been fully informed on the nature and interest to investigated radiosensitivity by the investigator.

Exclusion Criteria:

* No formal MMR meeting in the center where the patient has been treated
* No clinical and/or dosimetric available data
* No quality of life questionnaire completion whatever the cause
* Patients who do not agree to have at least one of the planed biologic tests, namely, skin biopsy and blood samples.
* Absence of affiliation to National French social security system
* Patient deprived of freedom or under legal protection (guardianship,curatorship)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-02 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Database of MMR boards | at 3 Months
  The PROUST national database of MMR boards, will be an opportunity to structure data collection on severe and durable radiation toxicity with an objective evaluation taking into account individual radiosensitivity.
Database of MMR boards | at 6 Months
  The PROUST national database of MMR boards, will be an opportunity to structure data collection on severe and durable radiation toxicity with an objective evaluation taking into account individual radiosensitivity.
Database of MMR boards | at 9 Months
  The PROUST national database of MMR boards, will be an opportunity to structure data collection on severe and durable radiation toxicity with an objective evaluation taking into account individual radiosensitivity.
Database of MMR boards | at 12 Months
  The PROUST national database of MMR boards, will be an opportunity to structure data collection on severe and durable radiation toxicity with an objective evaluation taking into account individual radiosensitivity.
Database of MMR boards | at 24 Months
  The PROUST national database of MMR boards, will be an opportunity to structure data collection on severe and durable radiation toxicity with an objective evaluation taking into account individual radiosensitivity.

SECONDARY OUTCOMES:
Radiation toxicity | at Day 0
  The rating scale NCI/CTCAE v4.03 will be used to differentiate between major and minor complications. Only major complications (grade > 3) will be included in the database.
Associated treatments to radiation | at Day 0, 3 Months, 6 Months, 9 Months,12 Months, 15 Months, 18 Months, 21 Months and 24 Months
  All drugs used either administered concurrently or sequentially with RT will be recorded
Follow-up and management strategy | at Day 0, 3 Months, 6 Months, 9 Months,12 Months, 15 Months, 18 Months, 21 Months and 24 Months
  Patients included in the database will have a planned follow-up every 3 to 6 months after inclusion during at least 2 years.The follow-up will be adjusted according to institution policy of the oncologic follow-up in case of regression of the clinical symptoms of toxicity.
Evolution of life's quality | at Day 0, 3 Months, 6 Months, 9 Months,12 Months, 15 Months, 18 Months, 21 Months and 24 Months
  The evaluation of the quality of life will be conducted using the Short-Form 36 questionnaire. This generic scale contains 36 items divided into eight dimensions, each corresponding to a different aspect of health and for a comprehensive assessment of the quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Yazid BELKACEMI, MD, PhD, Principal Investigator — Assistance Publique Hôpitaux de Paris (AP-HP)

IPD SHARING:
Plan to Share IPD: No
Datas are own by Assistance Publique - Hôpitaux de Paris, please contact sponsor for further information